CLINICAL TRIAL: NCT07222215
Title: A Phase II Multi-Center Open-label Randomized Study of CAPecitabine in Combination With ELAcestrant Versus Capecitabine Alone in Advanced Estrogen Receptor-Positive Breast Cancer (CAPELA)
Brief Title: PhII Randomized CAPecitabine + ELAcestrant vs. Capecitabine Alone in ER+ Breast Cancer (CAPELA)
Acronym: CAPELA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kristina A. Fanucci (Other)
Collaborators: Stemline Therapeutics, Inc. (Industry); Johns Hopkins University (Other); Translational Breast Cancer Research Consortium (Other); Menarini Group (Industry)
Responsible Party: Sponsor-Investigator, Kristina A. Fanucci, Sponsor-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25-605
Record Dates: First submitted 2025-10-23; First posted 2025-10-29 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Estrogen-receptor-positive Breast Cancer; Metastatic Breast Cancer; Breast Cancer; Hormone Receptor Positive Breast Cancer; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; HER2- Breast Cancer; ESR1 Gene Mutation; ER Wildtype; Breast Neoplasms
Keywords: Advanced Estrogen Receptor-Positive Breast Cancer; Metastatic Breast Cancer; Breast cancer; Hormone receptor positive breast cancer; Advanced Human Epidermal Growth Factor Receptor 2 negative breast cancer; HER2- Breast Cancer; ESR1 gene mutation; ER wildtype
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; elacestrant; RAD1901

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Capecitabine + Elacestrant (Experimental): Participants will be randomized 1:1, enrolled, and stratified based on the receipt of one or two prior lines of endocrine therapy in the metastatic setting, presence or absence of visceral disease, presence or absence of ESR1 mutation, and presence or absence of p53 mutation.
  * Baseline visit with assessments
  * Imaging every 9 weeks for 27 weeks, then every 12 weeks
  * Cycle 1 through End of Treatment (21-day cycles):
    * Days 1 - 14: Predetermined dose of Capecitabine 2x daily for 14 days followed by 7 days off
    * Days 1 - 21: Predetermined dose of Elacestrant 1x daily
  * Follow up: every 6 months after end of treatment
  Interventions: Drug: Capecitabine; Drug: Elacestrant
- Arm B: Capecitabine Monotherapy (Experimental): Participants will be randomized 1:1, enrolled, and stratified based on the receipt of one or two prior lines of endocrine therapy in the metastatic setting, presence or absence of visceral disease, presence or absence of ESR1 mutation, and presence or absence of p53 mutation.
  * Baseline visit with assessments
  * Imaging every 9 weeks for 27 weeks, then every 12 weeks
  * Cycle 1 through End of Treatment (21-day cycles):
    --Days 1 - 14: Predetermined dose of Capecitabine 2x daily for 14 days followed by 7 days off
  * Follow up: every 6 months after end of treatment
  Interventions: Drug: Capecitabine
- Optional switch after progression on Arm B Capecitabine monotherapy: Elacestrant Monotherapy (Experimental): For Arm B participants with ESR1 mutation, at the time of progression on Capecitabine participants have the option to continue on trial and switch to single agent Elacestrant monotherapy.
  -Imaging every 9 weeks for 27 weeks, then every 12 weeks
  Through End of Treatment (21-day cycles):
  --Days 1 - 21: Predetermined dose of Elacestrant 1x daily
  -Follow up: every 6 months after end of treatment
  Interventions: Drug: Elacestrant

INTERVENTIONS:
Drug: Capecitabine — A fluoropyrimidine carbamate, tablet taken orally, per standard of care.
  Other Names: Xeloda
  Arms: Arm A: Capecitabine + Elacestrant; Arm B: Capecitabine Monotherapy
Drug: Elacestrant — A selective estrogen receptor degrader, tablet taken orally, per standard of care
  Other Names: RAD1901; Elacestrant Dihydrochloride; RAD1901 - 2 HCl; C30H40Cl2N2O2
  Arms: Arm A: Capecitabine + Elacestrant; Optional switch after progression on Arm B Capecitabine monotherapy: Elacestrant Monotherapy

SUMMARY:
The goal of this research study is to compare a combination of two drugs, capecitabine and elacestrant to capecitabine alone as a treatment for advanced estrogen receptor-positive (ER+) breast cancer. This study is designed for participants with cancer that has previously stopped responding to medication in the class of therapy called CDK 4/6 inhibitors, including palbociclib, ribociclib, or abemaciclb.

The names of the study drugs involved in this study are:

* Elacestrant (a type of selective estrogen receptor degrader)
* Capecitabine (a type of fluoropyrimidine antimetabolite)

DETAILED DESCRIPTION:
This is a Phase II, multi-center, open-label, randomized study comparing a combination of two drugs, capecitabine and elacestrant, to capecitabine alone as a treatment for advanced estrogen receptor-positive (ER+) Human Epidermal Growth Factor Receptor 2 negative (HER2-) breast cancer. This study is designed for participants with cancer that has previously stopped responding to medication in the class of therapy called CDK 4/6 inhibitors, including palbociclib, ribociclib, or abemaciclb.

Participants will be randomized into one of two study groups: Arm A Capecitabine and Elacestrant versus Arm B Capecitabine alone. Randomization means a participants is placed into a study group by chance.

The U.S. Food and Drug Administration (FDA) has approved capecitabine as a treatment option for advanced estrogen receptor-positive (ER+) Human Epidermal Growth Factor Receptor 2 negative (HER2-) breast cancer.

The FDA has approved elacestrant for metastatic breast cancer with an ESR1 mutation. Elacestrant is not FDA approved for participants whose cancer does not have ESR1 mutation and it is possible elacestrant may not be as effective or effective at all in participants whose tumors do not have an ESR1 mutation.

The FDA has not approved Elacestrant and Capecitabine to be given together.

The research study procedures include screening for eligibility, in-clinic visits, questionnaires, blood tests, urine tests, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, and electrocardiograms (ECGs).

It is expected that about 297 people will take part in this research study.

Stemline, a Menarini Group Company, is supporting this research study by providing the study drugs, elacestrant, and funding. This study is also being supported by Johns Hopkins University on behalf of the Translational Breast Cancer Research Consortium (TBCRC).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed estrogen receptor-positive (ER+), HER2- negative metastatic or locally recurrent unresectable (advanced) invasive breast cancer.

ER and HER2 measurements should be performed according to institutional guidelines in a CLIA-approved setting. ER must be ≥ 10% on the most recent biopsy in which receptor testing was performed. Cutoff values for positive/negative HER2 staining should be in accordance with current ASCO/CAP (American Society of Clinical Oncology/College of American Pathologists) guidelines

* Participants must have standard of care testing documenting ESR1 mutation status. In patients without ESR1 mutation, this result must be from within 2 months.

  * qualifying ESR1 mutations: E380Q, V422del, S436P, L536H, L536P, L536R, Y537C, Y537D, Y537N, Y537S, D538G
* Women or men age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of capecitabine in combination with elacestrant participants <18 years of age are excluded from this study
* Women must be postmenopausal, which is defined as any of the following:

  * Age ≥ 60 years
  * Age < 60 and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression) and FSH and estradiol in the postmenopausal range per local normal range
  * Premenopausal women who have been on a GnRH agonist for at least three consecutive months prior to study entry are eligible. Women in this group MUST remain on the GnRH agonist for the duration of protocol treatment.
  * Status-post bilateral oophorectomy or total hysterectomy after adequate healing post-surgery
* Must have measurable or evaluable disease by RECIST 1.1. Must have progressed on at least one line of endocrine therapy in the metastatic setting or recurred on or within one year of adjuvant endocrine therapy
* Up to two prior endocrine therapies (with or without targeted treatment) are allowed in the advanced disease setting. If a patient recurred on or within one year of adjuvant endocrine therapy, it would be counted as one line of treatment.
* Prior CDK4/6 inhibition is required (in adjuvant or metastatic disease), unless a CDK4/6 inhibitor is contraindicated (CDK4/6 inhibitor in combination with endocrine treatment is considered as one line of endocrine treatment).
* Participants must have remained on a prior endocrine treatment alone or in combination with a CDK4/6 inhibitor in the metastatic setting without progression for at least 6 months prior to study entry. This regimen does not need to be the most recent regimen prior to study entry. If patients have progressed on adjuvant endocrine treatment and have not received treatment in the metastatic setting, they must have progressed after at least two years of adjuvant endocrine treatments.
* Prior alpelisib with endocrine treatment is allowed (considered as a line of endocrine treatment).
* Prior everolimus with endocrine treatment is allowed (considered a line of endocrine treatment).
* Prior capivasertib with endocrine treatment is allowed (considered a line of endocrine treatment)
* Prior fulvestrant is permitted. Prior elacestrant is NOT permitted, but prior other oral SERD is permitted.
* No prior chemotherapy regimen is allowed in the metastatic setting.
* Participants may have received radiotherapy for palliative purposes but must not be experiencing grade >1 treatment-related toxicities at study entry and must have completed treatment > 14 days prior to registration.
* ECOG PS 0-1
* Adequate hematological, liver, and kidney function, as defined below:

  * Absolute neutrophil count > 1,500/µL
  * Platelets > 100,000/µL
  * Hemoglobin > 9 g/dL (transfusion is allowed to meet this criterion) Total bilirubin < 1.5 x institutional upper limit or normal (ULN) or < 3 institutional ULN in the presence of documented Gilbert's syndrome
  * AST (SGOT)/ALT (SGPT) < 2.5 x institutional ULN, or ≤ 5 institutional ULN for subjects with documented metastatic disease to the liver
  * Creatinine clearance > 30 mL/min/1.73 m2 for subjects with creatinine levels above institutional ULN
* Women of childbearing age, women who are made postmenopausal through use of GNRH agonists, and men must agree to use adequate contraception for the duration of protocol treatment and for at least 6 months after the last dose of capecitabine.
* Premenopausal women must have a negative serum or urine pregnancy test. Pregnancy testing does not need to be pursued in female participants who are:

  * Age > 60 years; or
  * Age < 60 with intact uterus and amenorrhea for 12 consecutive months or more AND estrogen (estradiol) and FSH levels are within postmenopausal range; or
  * Status-post bilateral oophorectomy, total hysterectomy, or bilateral tubal ligation
* Participants must be able to swallow and retain oral medication.
* Ability to understand and the willingness to sign a written informed consent document.
* HIV-infected participants must have well-controlled HIV on ART, defined as:

  1. Participants on ART must have a CD4+ T-cell count ≥350 cells/mm3 at the time of screening.
  2. Participants on ART must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 or the LLOQ (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks before screening.
  3. It is advised that participants must not have had any AIDS-defining opportunistic infections within the past 12 months.
  4. Participants on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks before study entry (Day 1) and agree to continue ART throughout the study. The combination ART regimen must not contain any antiretroviral medications that interact with CYP3A4 inhibitors/inducers/substrates.

Note: No HIV testing is required at screening unless mandated by local health Authority.

* Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks, and have undetectable HBV viral load before allocation.

Note: Participants should remain on antiviral therapy throughout study intervention and follow local guidelines for HBV antiviral therapy post completion of study intervention.

Hepatitis B screening tests are not required unless:

* Known history of HBV infection
* As mandated by local health authority Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening. Note: Participants must have completed curative antiviral therapy at least 4 weeks before allocation.

Hepatitis C screening tests are not required unless:

* Known history of HCV infection
* As mandated by local health authority

Exclusion Criteria:

* Participants who have had endocrine and/or biologic therapy < 14 days prior to entering the study or those who have not recovered from any prior treatment-related toxicities (must recover to no more than grade 1; alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 toxicity not constituting a safety risk based on investigator's judgment are acceptable). This is to minimize risk of drug-drug interactions and clarify etiology of future toxicities.
* Participants who are receiving concurrent therapy with other investigational agents. This is to minimize risk of drug-drug interactions and clarify etiology of future toxicities.
* Rapidly progressive, symptomatic, visceral spread of disease placing participant at risk of life- threatening complications in the short term. It is likely that these patients will not benefit from this regimen.
* History of dihydropyrimidine dehydrogenase (DPD) deficiency. Patients with this deficiency are prone to significant toxicity from capecitabine.
* Participants with active brain metastases. Treated brain metastases that are asymptomatic and do not require systemic steroids for management of symptoms are allowed if they have received SRS (7-day washout) or WBRT (14-day washout) or asymptomatic untreated brain metastases measuring <1cm. Patients with leptomeningeal disease are not eligible. It is unlikely that these patients will benefit from this regimen.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection requiring systemic therapy, clinically significant cardiovascular disease including: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication, uncontrolled diabetes mellitus, gastrointestinal disorders potentially affecting the absorption of elacestrant, inflammatory bowel disease or chronic diarrhea, short bowel syndrome, or total gastric resection, or psychiatric illness/social situations that would limit compliance with study requirements. Active hepatitis B or active hepatitis C infection. Ability to comply with study requirements is to be assessed by each investigator at the time of screening for study participation. This could increase risk of toxicity from treatment and potentially decrease adherence to study protocol.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: (1) Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. (2) Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: ductal carcinoma in situ of the breast, cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin. History of prior malignancy puts patients at risk of recurrence from their prior malignancy or progression of a second malignancy which would complicate interpretation of the end points of this trial.
* Ongoing treatment with drugs that are sensitive substrates of P-glycoprotein (dabigatran, digoxin, fexofenadine) or BRCP (rosuvastatin, sulfasalazine). These drugs have potential drug-drug interactions with the study agents.
* Treatment with strong CYP3A inhibitors within 2 weeks before first study treatment administration or five elimination half-lives, whichever is longest and cannot be replaced.
* Medical conditions requiring concomitant administration of medications with a narrow therapeutic window metabolized by CYP3A and for which a dose reduction cannot be considered. See Appendix D for a list of medications that are CYP3A substrates. These drugs have potential drug-drug interactions with the study agents.
* Female participants lactating or nursing. The safety of these medications in pregnancy or breast feeding patients is unknown.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) in ESR1 mutant population | Tumor measurements are repeated every 3 cycles (each cycle is 21 days) for the first 9 cycles. After cycle 9 tumor measurements will be performed every 4 cycles.
  PFS based on the Kaplan-Meier method is defined as the time from study randomization to disease progression per RECIST 1.1 or death. Patients alive without disease progression are censored at the date of last disease evaluation.
Progression Free Survival (PFS) in intention to treat (ITT) population | Tumor measurements are repeated every 3 cycles (each cycle is 21 days) for the first 9 cycles. After cycle 9 tumor measurements will be performed every 4 cycles.
  PFS based on the Kaplan-Meier method is defined as the time from study randomization to disease progression per RECIST 1.1 or death. Patients alive without disease progression are censored at the date of last disease evaluation.

SECONDARY OUTCOMES:
Overall Survival (OS) in ESR1 mutant population | Follow up or other contact every 2 months for 24 months until time of second progression, then every 6 months for 5 years
  Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from randomization to death due to any cause or censored at date last known alive.
Objective Response Rate in ESR1 mutant population | Tumor measurements are repeated every 3 cycles (each cycle is 21 days) for the first 9 cycles. After cycle 9 tumor measurements will be performed every 4 cycles
  The objective response rate is defined as the rate of patients with a complete response or partial response, calculated using RECIST 1.1. The best overall response is the best response recorded from the start of treatment until disease progression/recurrence.
Clinical benefit rate (CBR) in ESR1 mutant population | Tumor measurements are repeated every 3 cycles (each cycle is 21 days) for the first 9 cycles. After cycle 9 tumor measurements will be performed every 4 cycles
  The clinical benefit rate is defined as the rate of patients with a complete response (CR), partial response (PR), or stable disease (SD) ≥24 weeks, calculated using RECIST 1.1.
Second progression event (PFS2) in ESR1 mutant population | Follow up or other contact every 2 months for a total of 24 months or until progressive disease
  PFS2 based on the Kaplan-Meier method is defined as the time from study randomization to second disease progression, according to RECIST 1.1, or death after first progression.
Overall survival (OS) in ITT population | Follow up or other contact every 2 months for 24 months until time of second progression, then every 6 months for 5 years
  Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from randomization to death due to any cause or censored at date last known alive.
Objective Response Rate in ITT population | Tumor measurements are repeated every 3 cycles (each cycle is 21 days) for the first 9 cycles. After cycle 9 tumor measurements will be performed every 4 cycles
  The objective response rate is defined as the rate of patients with a complete response or partial response, calculated using RECIST 1.1.
Clinical benefit rate (CBR) in ITT population | Tumor measurements are repeated every 3 cycles (each cycle is 21 days) for the first 9 cycles. After cycle 9 tumor measurements will be performed every 4 cycles
  The clinical benefit rate is defined as the rate of patients with a complete response (CR), partial response (PR), or stable disease (SD) ≥24 weeks, calculated using RECIST 1.1.
Second progression event (PFS2) in ITT population | Follow up or other contact every 2 months for a total of 24 months or until progressive disease
  PFS2 based on the Kaplan-Meier method is defined as the time from study randomization to second disease progression, according to RECIST 1.1, or death after first progression.
Safety and tolerability of capecitabine in combination with elacestrant | Assessment will occur once per cycle (each cycle is 21 days) for the first 9 cycles, then once every other cycle starting with cycle 10
  Assessment of toxicities and lab values categorized and graded according to CTCAE v5.0
Impact of treatment with capecitabine plus elacestrant versus capecitabine alone on quality of life | Once every 2 cycles (each cycle is 21 days) for the first 4 cycles, every 3 months for months 3-12 on trial, then every 6 months for months 12+ on trial
  evaluation with PRO-CTCAE and FACT-ES survey instruments

OTHER OUTCOMES:
Overall survival (OS) ESR1 mutation not detected population | Follow up or other contact every 2 months for 24 months until time of second progression, then every 6 months for 5 years
  Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from randomization to death due to any cause or censored at date last known alive.
Progression-free survival rate (PFS) | Tumor measurements are repeated every 3 cycles (each cycle is 21 days) for the first 9 cycles. After cycle 9 tumor measurements will be performed every 4 cycles
  PFS based on the Kaplan-Meier method is defined as the time from study randomization to disease progression per RECIST 1.1 or death. Patients alive without disease progression are censored at the date of last disease evaluation.
Second progression event (PFS2) | Follow up or other contact every 2 months for a total of 24 months or until progressive disease
  PFS2 based on the Kaplan-Meier method is defined as the time from study randomization to second disease progression, according to RECIST 1.1, or death after first progression.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Fanucci, MD, MHS, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States